CLINICAL TRIAL: NCT01716039
Title: A Study to Evaluate the Pharmacokinetics of Adalimumab in Combination With Methotrexate for the Treatment of Patients With Ulcerative Colitis
Brief Title: Pharmacokinetics of Adalimumab With Methotrexate for Treatment of Patients With Ulcerative Colitis (UC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to achieve recruitment target.
Sponsor: Alimentiv Inc. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RP1204
Record Dates: First submitted 2012-10-15; First posted 2012-10-29 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
Keywords: Moderately to severely active Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MTX 12.5 (Active Comparator): Receive once weekly oral dosing with MTX 12.5 mg (n=40) two weeks prior to the initiation of adalimumab 18 weekly doses of MTX and/or placebo in addition to doses of adalimumab
  Interventions: Drug: MTX 12.5; Drug: Adalimumab
- MTX 25 mg (Active Comparator): Once weekly oral dosing with MTX 25 mg (n=40) two weeks prior to the initiation of adalimumab 18 weekly doses of MTX in addition to doses of adalimumab
  Interventions: Drug: MTX 25; Drug: Adalimumab
- Placebo (Placebo Comparator): Once weekly oral dosing with placebo (n=20) two weeks prior to the initiation of adalimumab. Subjects will receive 18 weekly doses of placebo in addition to doses of adalimumab
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: MTX 12.5 — once weekly oral dosing with MTX 12.5 mg (n=40) two weeks prior to the initiation of adalimumab. Randomization will be stratified by disease activity (modified Mayo Score ≤9 or >9).
  Subjects will receive 18 weekly doses of MTX in addition to doses of adalimumab
  Other Names: MTX
  Arms: MTX 12.5
Drug: MTX 25 — once weekly oral dosing with MTX 25 mg (n=40) two weeks prior to the initiation of adalimumab. Randomization will be stratified by disease activity (modified Mayo Score ≤9 or >9).
  Subjects will receive 18 weekly doses of MTX in addition to doses of adalimumab
  Other Names: MTX
  Arms: MTX 25 mg
Drug: Adalimumab — Subjects will receive 18 weekly doses of adalimumab
  Other Names: Humira

SUMMARY:
Assess the body's reaction to dose-response relationship for the adalimumab/Methotrexate interaction in subjects with moderately to severely active ulcerative colitis.

DETAILED DESCRIPTION:
Assess the Pharmacokinetic dose-response relationship for the adalimumab/Methotrexate interaction in subjects with moderately to severely active UC.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females. Females of child bearing potential must have a negative serum pregnancy test prior to randomization, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
* Diagnosis of UC confirmed by established criteria, regardless of disease duration.
* Moderate to severely active UC, defined by a modified Mayo Score ≥6, with confirmed endoscopic activity by central reader (Mayo endoscopic subscore ≥2).
* Require initiation with adalimumab for induction of remission.
* Ability of subject to swallow study drug capsules.
* Ability of subject to participate fully in all aspects of this clinical trial.
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* Prior treatment with a TNF antagonist or biological therapy.
* Prior treatment with MTX.
* Disease limited to the rectum (proctitis).
* Documented presence of antibodies against adalimumab.
* Contraindication for anti-TNF or MTX therapy.
* Contraindication for endoscopy.
* Ostomy.
* Planned surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07-18 (Actual); Study Completion 2016-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feagan, MD, Principal Investigator — Robarts Research Institute - Western University

REFERENCES:
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Rutgeerts P, Van Assche G, Sandborn WJ, Wolf DC, Geboes K, Colombel JF, Reinisch W; EXTEND Investigators; Kumar A, Lazar A, Camez A, Lomax KG, Pollack PF, D'Haens G. Adalimumab induces and maintains mucosal healing in patients with Crohn's disease: data from the EXTEND trial. Gastroenterology. 2012 May;142(5):1102-1111.e2. doi: 10.1053/j.gastro.2012.01.035. Epub 2012 Feb 8. PMID 22326435
- [Background] Reinisch W, Sandborn WJ, Hommes DW, D'Haens G, Hanauer S, Schreiber S, Panaccione R, Fedorak RN, Tighe MB, Huang B, Kampman W, Lazar A, Thakkar R. Adalimumab for induction of clinical remission in moderately to severely active ulcerative colitis: results of a randomised controlled trial. Gut. 2011 Jun;60(6):780-7. doi: 10.1136/gut.2010.221127. Epub 2011 Jan 5. PMID 21209123
- [Background] Baert F, Noman M, Vermeire S, Van Assche G, D' Haens G, Carbonez A, Rutgeerts P. Influence of immunogenicity on the long-term efficacy of infliximab in Crohn's disease. N Engl J Med. 2003 Feb 13;348(7):601-8. doi: 10.1056/NEJMoa020888. PMID 12584368

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants randomized to receive placebo at Week 0 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks
  Adalimumab: 18 weekly doses of adalimumab
- MTX 12.5 mg: Participants randomized to receive Methotrexate 12.5 mg at Week 0 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks
  Adalimumab: 18 weekly doses of adalimumab
- MTX 25 mg: Participants randomized to receive Methotrexate 25.0 mg at Week 0 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks
  Adalimumab: 18 weekly doses of adalimumab
Period: Overall Study
Arm/Group | Placebo | MTX 12.5 mg | MTX 25 mg
Started | 4 | 8 | 10
Completed | 3 | 6 | 8
Not Completed | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- MTX 12.5 mg: Participants randomized to receive Methotrexate 12.5 mg at Week 0 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks
  Adalimumab:18 weekly doses of adalimumab
- MTX 25 mg: Participants randomized to receive Methotrexate 25.0 mg at Week 00 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks
  Adalimumab: 18 weekly doses of adalimumab
- Total: Total of all reporting groups
Arm/Group | Placebo | MTX 12.5 mg | MTX 25 mg | Total
Number analyzed (Participants) | 4 | 8 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.6) | 46.2 (13.7) | 48.5 (13.5) | 46.5 (13.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 3 | 7 | 14
  Female | 0 | 5 | 3 | 8
Disease Duration (Years) [Mean (Standard Deviation); unit: years] | 10.8 (8.0) | 5.1 (3.7) | 7.0 (9.3) | 7.0 (7.4)
Weight [Mean (Standard Deviation); unit: kg] | 75.0 (15.3) | 75.5 (15.2) | 89.6 (20.5) | 81.8 (18.5)
C-Reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] | 6.6 (3.9) | 5.2 (2.7) | 15.1 (16.1) | 9.9 (11.8)
Fecal Calprotectin [Mean (Standard Deviation); unit: ug/g] | 606.7 (566.6) | 675.8 (431.6) | 545.2 (362.0) | 603.7 (400.1)
Mayo Clinic Score [Mean (Standard Deviation); unit: units on a scale] — The Mayo Clinic Score includes 4 variables: stool frequency, rectal bleeding, a physician's global assessment, and endoscopic findings with flexible sigmoidoscopy. Each variable is scored on a 4-point scale (0-3 points) and summed to give a total disease activity score (maximum score = 12), with higher scores representing more severe disease activity
  units on a scale | 9.0 (1.2) | 8.6 (2.1) | 8.7 (2.1) | 8.7 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Modified Baron Score From Baseline to the Final Visit (Week 18) Between the Treatment Groups
Description: The modified Baron score is scored on a 0-4 scale that evaluates friability, vascular pattern, bleeding and ulceration on a 5-point grading scale with a higher score indicating more severe disease activity.
  The mean change and 95% CI are based on least square means from the analysis of covariance
Time Frame: Baseline up to Week 18
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants randomized to receive placebo at Week 0 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks.
  Adalimumab: 18 weekly doses of adalimumab
- MTX 12.5mg: Participants randomized to receive Methotrexate 12.5 mg at Week 0 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks.
  Adalimumab: 18 weekly doses of adalimumab
Arm/Group | Placebo | MTX 12.5mg | MTX 25 mg
Number analyzed (Participants) | 4 | 8 | 10
score on a scale | 0.7 (1.2) | 1.1 (1.6) | 0.9 (1.8)
Statistical Analysis 1: Comparison: Placebo vs MTX 12.5mg; Test type: Other — Comparing the change in the modified Baron score from baseline to week 18 between the treatment groups; p = 0.758, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs MTX 25 mg; Test type: Other; p = 1.00, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in the Ulcerative Colitis Endoscopic Index of Severity (UCEIS) Score From Baseline to the Final Visit (Week 18) Between the Treatment Groups.
Description: UCEIS is a simple scoring tool that contains3 items (vascular pattern, bleeding, and ulceration).
  The UCEIS scores 3 endoscopic items: vascular pattern (ranges 0-2 points), bleeding (ranges 0-3 points), and the presence of ulcers and erosions (ranges 0-3 points).The total UCEIS is calculated by adding up the 3 item scores(range,0-8points), with higher scores representing more severe disease activity.
  The mean change and 95% CI are based on least square means from the analysis of covariance
Time Frame: Baseline up to Week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- MTX 25 mg: Participants randomized to receive Methotrexate 25.0 mg at Week 0(two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks
  Adalimumab: 18 weekly doses of adalimumab
Arm/Group | Placebo | MTX 12.5 mg | MTX 25 mg
Number analyzed (Participants) | 4 | 8 | 10
score on a scale | 0.5 [-2.3 to 3.4] | 0.7 [-1.0 to 2.4] | 1.1 [-0.6 to 2.7]
Statistical Analysis 1: Comparison: Placebo vs MTX 12.5 mg vs MTX 25 mg; Test type: Other; p = 0.908, ANCOVA — p-value for the overall treatment difference is based on an analysis of covariance adjusting for baseline UCEIS

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 18 weeks
Groups:
- MTX 25 mg: Participants randomized to receive Methotrexate 25.0 mg at Week 00 (two weeks prior to the initiation of adalimumab induction therapy) and then every week for 18 weeks
  Adalimumab:18 weekly doses of adalimumab
Arm/Group | Placebo | MTX 12.5 mg | MTX 25 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/8 | 1/10
Other Adverse Events (participants affected / at risk) | 3/4 | 8/8 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | MTX 12.5 mg (N=8) | MTX 25 mg (N=10)
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | MTX 12.5 mg (N=8) | MTX 25 mg (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1 | 0
Dysgeusia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Contusion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Throat irritation (Gastrointestinal disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI of this Investigator-Initiated study had right to prior publication. If PI did not commence publication within 12months after the close of trial at all sites or after PI's manuscript was accepted for publication, whichever occurs first, the Sub-I and Sub-Institution were free to publish or present, provided that the Sub-I provided to the PI any doc. to be submitted for publication at least 30days prior to the planned date of submission for publication to permit a review of the Manuscript.